CLINICAL TRIAL: NCT00149786
Title: Treatment of Adolescents With Anorexia Nervosa
Brief Title: Effectiveness of Family-Based Versus Individual Psychotherapy in Treating Adolescents With Anorexia Nervosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH070621 (NIH); R01MH070621 (NIH); DDTR B4-ARE
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Eating Disorders
Keywords: Anorexia Nervosa; Adolescents; Family therapy; Individual therapy
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Those adolescents receiving family based therapy
  Interventions: Behavioral: Family Based Therapy
- 2 (Active Comparator): Those adolescents receiving individual therapy
  Interventions: Behavioral: Ego-Oriented Individual Psychotherapy

INTERVENTIONS:
Behavioral: Family Based Therapy — Family therapy will be given for a total of 24 hours over the course of 12 months.
  Other Names: FBT
  Arms: 1
Behavioral: Ego-Oriented Individual Psychotherapy — Individual therapy will be given for a total of 24 hours over the course of 12 months.
  Other Names: EOIP
  Arms: 2

SUMMARY:
This study will compare the effectiveness of family-based therapy versus individual psychotherapy for the treatment of adolescent anorexia nervosa.

DETAILED DESCRIPTION:
In adolescents, anorexia nervosa severely affects physical, emotional, and social development. Despite the seriousness and prevalence of adolescent anorexia nervosa, few studies have focused on the effectiveness of various types of psychotherapy treatment. Family-based therapy may be an effective approach to treating adolescent anorexia nervosa. This study will compare the effectiveness of family-based therapy versus ego-oriented individual psychotherapy for the treatment of adolescent anorexia nervosa. Simultaneously, it will examine potential predictors, mediators, and moderators of weight gain, psychological concerns about weight and shape, and changes in family functioning.

Participants in this open-label study will be randomly assigned to receive one of two types of therapy: family-based therapy or ego-oriented individual psychotherapy. Both types of therapy will be given for a total of 24 hours over the course of 12 months. Physical and psychological assessments will be completed during study visits at baseline, immediately post-treatment, six months post-treatment, and one year post-treatment. Amount of weight gain will be evaluated, along with changes in weight and body shape concerns, as measured by the Eating Disorder Examination.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for anorexia nervosa
* Lives with at least one parent who is willing to participate
* Medically stable
* Adequate transportation to clinic
* Proficient at speaking, reading, and writing English

Exclusion Criteria:

* Currently undergoing treatment or taking medication that may affect eating or weight

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Scores on the Eating Disorders Examination | Measured at Year 1 of treatment and Year 1 of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: James D. Lock, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- The University of Chicago, Pritzker School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Le Grange D, Lock J, Accurso EC, Agras WS, Darcy A, Forsberg S, Bryson SW. Relapse from remission at two- to four-year follow-up in two treatments for adolescent anorexia nervosa. J Am Acad Child Adolesc Psychiatry. 2014 Nov;53(11):1162-7. doi: 10.1016/j.jaac.2014.07.014. Epub 2014 Aug 23. PMID 25440306
- [Derived] Lock J, Le Grange D, Agras WS, Moye A, Bryson SW, Jo B. Randomized clinical trial comparing family-based treatment with adolescent-focused individual therapy for adolescents with anorexia nervosa. Arch Gen Psychiatry. 2010 Oct;67(10):1025-32. doi: 10.1001/archgenpsychiatry.2010.128. PMID 20921118